CLINICAL TRIAL: NCT04823026
Title: Host RNA Profiles to Detect Infections in Young Infants
Acronym: CHILD_YIC
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kia Hee Schultz Dungu, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: H-18065635-YIC
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Bacterial Infections; Urinary Tract Infections; Sepsis; Fever; Viral Infection; Infant, Newborn, Disease; Bacteremia; Meningitis
MeSH Terms: conditions — Bacterial Infections; Urinary Tract Infections; Sepsis; Fever; Virus Diseases; Disease; Bacteremia; Meningitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All included young infants will have 0.50 - 2.50 ml whole blood drawn into PAXgene blood RNA tubes (Qiagen®) along with routine blood tests within 48 hours of admission. Host RNA expression profiling (whole transcriptome profiling) by RNA sequencing will be performed at the Centre for Genomic Medicine, Rigshospitalet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: 70 young infants with proven bacterial infection.
  Interventions:
  Diagnostic test: Host RNA expression profiling (whole transcriptome profiling) using whole blood RNA sequencing. Cases will be randomly assigned to a "Discovery Cohort" (identification of diagnostic RNA profiles) or a "Validation Cohort" (validation of the identified RNA profiles).
- Group 2: 70 young infants with non-bacterial infection.
  Interventions:
  Diagnostic test: Host RNA expression profiling (whole transcriptome profiling) using whole blood RNA sequencing. Cases will be randomly assigned to a "Discovery Cohort" (identification of diagnostic RNA profiles) or a "Validation Cohort" (validation of the identified RNA profiles).
- Group 3: 30 young infants without infection.
  Interventions:
  Diagnostic test: Host RNA expression profiling (whole transcriptome profiling) using whole blood RNA sequencing. Cases will be randomly assigned to a "Discovery Cohort" (identification of diagnostic RNA profiles) or a "Validation Cohort" (validation of the identified RNA profiles).

SUMMARY:
This study seeks to identify and test host RNA expression profiles as markers for infections in young infants. Preliminary studies have shown high sensitivity and specificity for the discrimination of bacterial from non-bacterial infections in children, but the method has only been investigated in a limited number of young infants. The study aims to include 65 young infants with serious bacterial infections. The samples will be analysed by RNA sequencing. New diagnostic tools may help reduce unnecessary antibiotic treatment, antibiotic resistance, side-effects, hospitalisation and invasive procedures.

DETAILED DESCRIPTION:
Background:

Infections in young infants is a challenge as 1) it is often not possible to distinguish serious bacterial infection (SBI) from viral infection by clinical appearance alone, 2) a causative organism is often not identified and 3) due to relatively low sensitivity and specificity of current biomarkers. The consequence is overtreatment with antibiotics being prescribed to as many as 50% of febrile young infants presenting to emergency departments. However, the majority of these children does not have a bacterial infection. Host RNA expression profiling has shown high sensitivity and specificity for discriminating bacterial from non-bacterial infections in preliminary studies of febrile young infants.

Methods:

A prospective multicentre observational study including young infants admitted and evaluated due to suspected infection at the 4 paediatric acute care units in the Capital Region of Denmark (Rigshospitalet, Hvidovre Hospital, Herlev Hospital, Nordsjællands Hospital - Hillerød). Whole blood will be collected in PAXgene blood RNA tubes and analysed by RNA sequencing at the Centre for Genomic Medicine, Rigshospitalet. Host RNA expression profiles will be identified in a discovery cohort and the diagnostic performance will be tested in a validation cohort. A control group of healthy and afebrile young infants will be included.

Time frames:

Patient recruiting: May 15th 2020 to February 28th 2022. Sample analysis (RNA sequencing): March 1st 2022 to August 31st 2022.

Perspectives:

New molecular-based diagnostic tools complementary to conventional methods may optimise infection management in young infants by improving early diagnostics and allowing early modification of antibiotic treatment. This will reduce antibiotic resistance, side effects, unnecessary hospitalisation and invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

1. age 0-3 months
2. admitted from home
3. suspected of infection
4. having routine blood sampling done
5. gestational age or corrected gestational age greater than or equal to 37+0
6. informed consent

Exclusion Criteria:

1. not possible to draw blood tests
2. withdrawal of consent
3. sampling >48 hours after admission

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young infants suspected of infection and admitted to one of the 4 paediatric departments in the Capital Region of Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Host RNA expression profiles | 21 months
  To identify specific host RNA expression profiles in whole blood in response to bacterial infections in young infants

SECONDARY OUTCOMES:
Application of known host RNA profiles | 21 months
  To test host RNA profiles published in other studies, e.g. based on the genes IFI44L and FAM89A
Time study | 21 months
  To investigate the change in host RNA expression over time during an infection period

CONTACTS AND LOCATIONS:
Overall Officials: Kia Hee Schultz Dungu, MD, Principal Investigator — Rigshospitalet, Denmark; Ulrikka Nygaard, Ass Prof PhD, Study Chair — Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Department of Paediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen
  - Department of Paediatrics and Adolescent Medicine, Herlev Hospital, Herlev
  - Department of Paediatrics and Adolescent Medicine, Nordsjællands Hospital - Hillerød, Hillerød
  - Department of Paediatrics, Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: Undecided